CLINICAL TRIAL: NCT00948714
Title: Peer and Health Educator Support for Cardiovascular Health in African-American Primary Care Patients
Brief Title: Support for Cardiovascular Health in African American Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 808214
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Diseases; Blood Pressure
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case (Experimental)
  Interventions: Behavioral: Peer Coach Phone Calls; Behavioral: Health Educator Visits; Other: written materials
- Control (Active Comparator)
  Interventions: Other: written materials

INTERVENTIONS:
Behavioral: Peer Coach Phone Calls — Subjects will receive 3 phone calls from a trained peer coach over 6 months.
  Arms: Case
Behavioral: Health Educator Visits — Subjects will meet 2 times with a trained health educator in the practice
  Arms: Case
Other: written materials — Subjects will receive written material and brochures and a cookbook from the American Heart Association addressing healthy lifestyle

SUMMARY:
Project Overview:

Poor hypertension control has dire consequences for the African-American population who suffer greater death and disability from heart disease, stroke, and renal failure than whites. To reduce these health disparities it is critical to promote of a healthy lifestyle in regard to diet, exercise, adherence to medications, as well as other behaviors. However, physicians usually fail to address lifestyle behaviors in the context of the harried patient visit. Therefore, the investigators hypothesized that the investigators could reduce cardiovascular risk by providing additional support to persons with poorly controlled hypertension through phone calls from trained peer patients and visits to an office support staff member.

Study Design:

A single-blind, randomized, controlled trial in 280 African-American primary care patients aged 40-75 with poorly controlled hypertension (HTN). The intervention group receives a practice-based team intervention that combines peer coach with office staff (i.e., medical assistant or licensed practice nurse) visits to address lifestyle challenges. Both intervention and control groups receive informational materials and healthy soul food recipes from the American Heart Association. The 6 month intervention alternates monthly phone calls from peer coaches about lifestyle behavioral changes with office-based visits with the support staff member during which patients review and discuss low literacy slide shows about healthy behaviors as well as examine their personal cardiovascular risk profile.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Uncontrolled Hypertension
* at least 3 practice visits in the past 2 years
* One lipid panel since 2005

Exclusion Criteria:

* No recent lipid panel
* Kept less than 60% of primary care visits in the prior 2 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Greater reduction in CHD risk in case group vs. control | 6 months

SECONDARY OUTCOMES:
5mm reduction in systolic blood pressure in case group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Weiner, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Edward S. Cooper Practice of General Internal Medicine, Philadelphia, Pennsylvania
  - PennCare Internal Medicine Associates, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Turner BJ, Hollenbeak CS, Liang Y, Pandit K, Joseph S, Weiner MG. A randomized trial of peer coach and office staff support to reduce coronary heart disease risk in African-Americans with uncontrolled hypertension. J Gen Intern Med. 2012 Oct;27(10):1258-64. doi: 10.1007/s11606-012-2095-4. Epub 2012 May 9. PMID 22570108